CLINICAL TRIAL: NCT02070978
Title: A Phase IIb, Multi-Center, Long-Term Extension Trial to Evaluate the Safety and Tolerability of Atacicept in Subjects With Systemic Lupus Erythematosus (SLE) Who Completed Protocol EMR-700461-023 (ADDRESS II)
Brief Title: Long-term Safety and Tolerability of Atacicept (Long-term Follow-Up of Participant Who Participated in ADDRESS II)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to shortage of drug supply.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 700461-024; 2013-002758-62 (EudraCT Number)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus Erythematosus, Systemic; Atacicept 75 and 150 mg; LTE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Atacicept 75 mg (Experimental)
  Interventions: Drug: Atacicept 75 mg
- Atacicept 150 mg (Experimental)
  Interventions: Drug: Atacicept 150 mg
- Placebo/Atacicept 150 mg (Experimental)
  Interventions: Drug: Atacicept 150 mg

INTERVENTIONS:
Drug: Atacicept 75 mg — Participants who received atacicept 75 milligram (mg) as once-weekly subcutaneous injection in the core study ADDRESS II continued to receive this dose during this LTE study. Participants in this reporting arm received the medication up to a maximum of 143.7 weeks.
  Arms: Atacicept 75 mg
Drug: Atacicept 150 mg — Participants who received placebo in the core study ADDRESS II switched to receive atacicept 150 mg as once-weekly subcutaneous injection for up to a maximum of 97.7 weeks during this LTE study.
  Arms: Placebo/Atacicept 150 mg
Drug: Atacicept 150 mg — Participants who received atacicept 150 mg in core study ADDRESS II continued to receive atacicept 150 mg as once-weekly subcutaneous injection during this LTE study up to a maximum of 97.9 weeks.
  Arms: Atacicept 150 mg

SUMMARY:
This is a multicenter, double-blind, Phase 2b, long-term extension (LTE) to the ADDRESS II core trial (EMR 700461-023) (NCT01972568), to evaluate long-term safety and tolerability of atacicept in participants with systemic lupus erythematosus (SLE). Participants who completed the 24-week core study ADDRESS II core study (NCT01972568) and thus not met any of the discontinuation criteria were invited to enter this long-term extension (LTE) study NCT02070978.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had completed the 24-week treatment period of study EMR-700461-023 (ADDRESS II core trial)
* Women of childbearing potential who had a negative pregnancy test
* Other protocol defined inclusion criteria were applied

Exclusion Criteria:

* Active neurological symptoms of SLE that were deemed severe or progressive
* Diagnosis of any demyelinating disease, such as, but not restricted to, multiple sclerosis (MS) or optic neuritis
* Pregnancy
* Active clinically significant viral, bacterial, or fungal infection, or any major episode of infection that in the investigator's opinion makes the participants unsuitable to continued participation in the study
* Other protocol defined exclusion criteria were applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (84):
- United States (23):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - University of Alabama at Birmingham - (UAB), Birmingham, Alabama
  - Wallace Rheumatic Study Center, Beverly Hills, California
  - Southern California Permenent Medical Group, Fontana, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Clinical Research of West Florida - Corporate, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - McIlwain Medical Group, PA, Tampa, Florida
  - AA MRC LLC Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Clayton Medical Associates, P.C., St Louis, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Hospital for Special Surgery, New York, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - MetroHealth System, Cleveland, Ohio
  - Arthritis & Rheumatology Center of Oklahoma, Oklahoma City, Oklahoma
  - OMRF, Oklahoma City, Oklahoma
  - Clinical Research Center of Reading LLC, Wyomissing, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Austin Regional Clinic, P.A., Austin, Texas
  - Little River Arthritis & Osteoporosis Clinic, Waco, Texas
- Argentina (10):
  - Instituto CAICI, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Centro Integral de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Organizacion Medica de Investigacion (OMI), Ciudad Autonoma Buenos Aires
  - APRILLUS, Ciudad Autonoma Buenos Aires
  - Atencion Integral en Reumatologia (AIR), Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Cordis S.A., Salta
  - Centro Polivalente de Asistencia e Inv. Clinica CER, San Juan
- Centro de Pesquisas em Diabetes Ltda., Porto Alegre, Rio Grande do Sul, Brazil
- Bulgaria (7):
  - MHAT "Eurohospital" - Plovdiv, OOD, Plovdiv
  - Medical Center "Teodora", EOOD, Rousse
  - MHAT - Ruse, AD, Rousse
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - DCC "Sveta Anna", EOOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - MHAT-Targovishte, AD, Targovishte
- Chile (6):
  - Corporacion de Beneficencia Osorno, Osorno
  - Quantum Research Santiago, Puerto Varas
  - Centro Medico Prosalud, Santiago
  - Biomedica, Santiago
  - Centro de Estudios Reumatologicos, Santiago
  - CINVEC - Centro de Investigacion Clinica V Region, Viña del Mar
- Czechia (2):
  - Revmatologicky Ustav, Prague
  - Revmatologicka ambulance, Uherské Hradiště
- Germany (2):
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
- Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan, Italy
- Mexico (9):
  - Hospital Universitario de Saltillo "Dr. Gonzalo Valdés Valdés", Saltillo, Coahuila
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Icle S.C., Guadalajara, Jalisco
  - Unidad de Investigacion en Enfermedades Cronico Degenerativas SC, Guadalajara, Jalisco
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Clinica de Enfermedades Cronicas y de Procedimientos Especiales, S.C., Morelia, Michoacán
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Centro Multidisciplinario para el desarrollo Especializado de la Investigacion Clinica en Yucatan, Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
- Peru (3):
  - Hogar Clínica San Juan de Dios - Arequipa, Arequipa
  - Clinica Medica Cayetano Heredia, Lima
  - Invest Clinicas Sac Inst de Ginecologia y Reproduccion, Lima
- Philippines (4):
  - Angeles University Foundation Medical Center, Angeles City, Pampanga
  - Mary Mediatrix Medical Center, Batangas
  - Davao Doctors Hospital, Davao City
  - Iloilo Doctors Hospital, Iloilo City
- Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz, Poland
- Russia (6):
  - FSBEI HE " First Moscow State Medical University n.a. I.M. Sechenov" of the MoH of the RF, Moscow
  - SBIH of Republic Kareliya "Republican Hospital n.a. V.A. Baranov", Petrozavodsk
  - SPb SBIH "Clinical Rheumatological Hospital # 25", Saint Petersburg
  - SIH "Saratov City Clinical Hospital # 12", Saratov
  - SBIH of Vladimir region "Regional Clinical Hospital", Vladimir
  - SBHI of Yaroslavl Region "Clinical Hospital # 8", Yaroslavl
- South Africa (2):
  - Naidoo, A, Durban, KwaZulu-Natal
  - Winelands Medical Research Centre, Stellenbosch, Western Cape
- South Korea (3):
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Konkuk University Medical Center, Seoul
- Hospital Clinico Universitario de Valladolid, Valladolid, Spain
- United Kingdom (3):
  - Queen's Hospital, Romford, Essex
  - University College London Hospitals, London, Greater London
  - Guy's Hospital, London, Greater London

REFERENCES:
- [Derived] Wallace DJ, Isenberg DA, Morand EF, Vazquez-Mateo C, Kao AH, Aydemir A, Pudota K, Ona V, Aranow C, Merrill JT. Safety and clinical activity of atacicept in the long-term extension of the phase 2b ADDRESS II study in systemic lupus erythematosus. Rheumatology (Oxford). 2021 Nov 3;60(11):5379-5389. doi: 10.1093/rheumatology/keab115. PMID 33547784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed 24-week of the ADDRESS II core study (NCT01972568) and didn't meet any discontinuation criteria were enrolled in this long-term extension (LTE) study NCT02070978. The study was conducted at 81 sites in 17 countries in Asia, Europe, North America, Central America, and South America.
Pre-assignment Details: Participants who received placebo in core study ADDRESS II were switched to receive atacicept 150 milligram (mg) as once-weekly subcutaneous injections in LTE study. Participants who received atacicept 75 mg or 150 mg in core study ADDRESS II continued to receive the respective randomized dosage as once-weekly subcutaneous injections in LTE study.
Groups:
- Placebo/Atacicept 150 mg: Participants received atacicept 150 mg as once-weekly subcutaneous injection during this LTE study up to a maximum of 97.7 weeks.
- Atacicept 75 mg: Participants received atacicept 75 mg as once-weekly subcutaneous injection during this LTE study up to a maximum of 143.7 weeks.
- Atacicept 150 mg: Participants received atacicept 150 mg as once-weekly subcutaneous injection during this LTE study up to a maximum of 97.9 weeks.
Period: Overall Study
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Started | 83 | 82 | 88
Completed | 36 | 29 | 35
Not Completed | 47 | 53 | 53
Not completed — Adverse Event | 6 | 2 | 0
Not completed — Lost to Follow-up | 1 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 5 | 3
Not completed — Protocol Violation | 1 | 0 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Death | 0 | 0 | 2
Not completed — Un-specified | 3 | 2 | 2
Not completed — Terminated by Sponsor | 33 | 40 | 39

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) analysis set: defined as all enrolled participants in the LTE study. Efficacy analyses were performed on the mITT analysis set according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg | Total
Number analyzed (Participants) | 83 | 82 | 88 | 253
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (13.0) | 37 (10.7) | 38 (11.5) | 39 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 75 | 82 | 231
  Male | 9 | 7 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 43 | 40 | 131
  Not Hispanic or Latino | 35 | 39 | 48 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 3 | 10
  Asian | 7 | 13 | 13 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 3 | 7 | 13
  White | 64 | 58 | 55 | 177
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Serious Adverse Event (SAE) During the Treatment Period
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. Treatment- Emergent adverse events (TEAEs) during the treatment period exclude those ongoing at the time of study entry into 024 LTE Day 1 and exclude the safety follow-up period.
Time Frame: Baseline (LTE Day 1) up to maximum treatment duration of 143.7 weeks
Population: The safety analyses set included all participants enrolled into the LTE study and who received at least 1 dose of planned study treatment. Participants were analyzed according to the actual treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Participants | 13 | 10 | 9

2. Primary Outcome: Number of Participants Who Prematurely Discontinued the Treatment Due to Adverse Event (AE)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. TEAEs were defined as events with an onset date on or after the date of first dose of study treatment in the core study and ongoing at the 024 LTE study entry, occurring during the 024 LTE study and the Safety follow-up Period.
Time Frame: Baseline (Day 1 of Core study) up to maximum duration of 167.7 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Participants | 9 | 4 | 5

3. Secondary Outcome: Change From Baseline in Systemic Lupus International Collaborating Clinics/American College of Rheumatology (SLICC/ACR) Damage Index Organ Damage Scores
Description: SLICC/ACR score or damage index evaluates cumulative damage in Systemic Lupus Erythematosus (SLE). These changes may or may not be related to SLE. Most items are scored only if they have been present for at least 6 months. Scores range from 0 to 47 points, with higher scores indicating greater cumulative damage. Baseline was defined as Day 1 of Core study.
Time Frame: Baseline: Day 1 (Core Study), Day 1 (LTE Study), Week 24, Week 48, Week 72 and Week 96
Population: Modified intent-to-treat (mITT) analysis set was defined as all enrolled participants in the LTE study. Efficacy analyses were performed on the mITT analysis set according to randomized treatment. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified categories.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Baseline; Day 1 (Core Study) | 1 (1.0) | 1 (1.2) | 0 (0.8)
  Change at LTE Day 1 | 0 (0.0) | 0 (0.1) | 0 (0.0)
  Change at LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  Change at LTE Week 24 | 0 (0.1) | 0 (0.1) | 0 (0.2)
  Change at LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  Change at LTE Week 48 | 0 (0.2) | 0 (0.2) | 0 (0.3)
  Change at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Change at LTE Week 72 | 0 (0.3) | 0 (0.3) | 0 (0.2)
  Change at LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  Change at LTE Week 96 | 0 (0.3) | 0 (0.3) | 0 (0.0)

4. Secondary Outcome: Change From Baseline in Disease Activity as Measured by British Isles Lupus Assessment Group (BILAG) 2004 Score
Description: BILAG Disease Activity Index evaluates systemic lupus erythematosus (SLE) activity in 8 organ system domains: General, mucocutaneous, neurological, musculoskeletal, cardiorespiratory, vasculitis, renal, and hematologic using a separate alphabetic score (A to E) assigned to each organ system defined as follows. BILAG A: Severe disease activity; BILAG B: moderate disease activity; BILAG C: mild disease; BILAG D: system previously affected but now inactive; BILAG E: system never involved. BILAG evaluated by scoring each of a list of signs and symptoms as: improving (1); same (2); worse (3); new (4); not present (0); not done (ND). The total BILAG score is the sum of the scores of the 8 domains where A=9, B=3, C=1, D=0, and E=0. The total score ranges from 0 to 72 with a higher score indicating greater lupus activity.
Time Frame: Baseline: Core study Screening, LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: mITT analysis set was defined as all enrolled participants in the LTE study. Efficacy analyses were performed on the mITT analysis set according to randomized treatment. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified categories.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Baseline: Core study Screening | 15 (7.1) | 14 (7.2) | 16 (6.1)
  Change at LTE Day 1 | -8 (6.9) | -9 (7.2) | -10 (6.8)
  Change at LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  Change at LTE Week 24 | -8 (8.3) | -10 (7.5) | -12 (7.2)
  Change at LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  Change at LTE Week 48 | -9 (7.7) | -8 (7.5) | -11 (7.4)
  Change at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Change at LTE Week 72 | -9 (7.9) | -10 (6.2) | -11 (8.2)
  Change at LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  Change at LTE Week 96 | -14 (12.9) | -8 (6.3) | -12 (6.8)

5. Secondary Outcome: Change From Baseline in Disease Activity as Measured by Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K) Score
Description: SLEDAI-2K is an activity index that measures disease activity and records feature of active lupus as present or not present. SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms). Baseline was defined as core study screening visit.
Time Frame: Baseline: Screening Visit (Core Study); LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: mITT analysis set was defined as all enrolled participants in the LTE study. Efficacy analyses were performed on the mITT analysis set according to randomized treatment. Here, "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified categories.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Baseline: Screening Visit (Core Study) | 10 (2.9) | 10 (3.4) | 10 (3.0)
  Change at LTE Day 1 | -4 (4.1) | -5 (4.5) | -5 (3.9)
  Change at LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  Change at LTE Week 24 | -5 (4.3) | -6 (4.1) | -6 (3.9)
  Change at LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  Change at LTE Week 48 | -6 (3.4) | -6 (4.6) | -7 (4.3)
  Change at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Change at LTE Week 72 | -5 (3.8) | -6 (3.7) | -7 (3.9)
  Change at LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  Change at LTE Week 96 | -7 (5.0) | -6 (4.9) | -8 (2.7)

6. Secondary Outcome: Change From Baseline in Disease Activity as Measured by SLEDAI-2K Responder Index-50 (SRI-50) Score
Description: SRI-50 index was derived from SLEDAI-2K and could capture 50% or better improvement in each descriptor between any 2 visits in systemic lupus erythematosus (SLE) participants when there was incomplete resolution. The new assigned scores for the descriptors of SRI-50 were derived by dividing the score of each SLEDAI-2K descriptor by 2. SLEDAI-2K was an activity index that measured disease activity and records feature of active lupus as present or not present. SLEDAI-2K used a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms. Each symptom present was assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranged from 0 points (no symptoms) to 105 points (presence of all defined symptoms).
Time Frame: Baseline: Screening Visit (Core Study); LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: Data was not collected for this endpoint as the results from ADDRESS II core study (700461-023; NCT01972568) for SRI-50 were not significant. Therefore, data collection for the SRI-50 for current study (700461-024; NCT02070978) was halted and no analysis was conducted for endpoint.
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Disease Activity as Measured by Physician's Global Assessment (PGA) Score
Description: The PGA was used to quantify disease activity and was measured using an anchored visual analog scale (VAS). The participant's current disease activity assessed by investigator in the score range of 0 to 3. Where 0=none; 1=mild; 2=moderate; 3=severe. The assessment made relative not to the participant's most severe state, but the most severe state of systemic lupus erythematosus (SLE) per the investigator's assessment. Baseline was defined as core study screening visit.
Time Frame: Baseline: Screening Visit (Core Study); LTE Day1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Baseline: Screening Visit (Core Study) | 1.56 (0.424) | 1.46 (0.509) | 1.47 (0.460)
  Change at LTE Day 1 | -0.76 (0.559) | -0.77 (0.559) | -0.77 (0.614)
  Change at LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  Change at LTE Week 24 | -0.91 (0.620) | -0.85 (0.555) | -0.94 (0.547)
  Change at LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  Change at LTE Week 48 | -1.01 (0.647) | -0.86 (0.522) | -0.99 (0.557)
  Change at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Change at LTE Week 72 | -0.90 (0.758) | -0.84 (0.503) | -1.03 (0.580)
  Change at LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  Change at LTE Week 96 | -1.17 (0.518) | -0.72 (0.579) | -1.21 (0.411)

8. Secondary Outcome: Number of Participants Who Achieved SLE Responder Index (SRI-4) Response (a Disease Activity Composite Index)
Description: SRI-4 response was defined as greater than or equal to 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score, no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score and no worsening (less than 10 percent increase) from baseline Physician's Global Assessment of Disease Activity (PGA). SLEDAI-2K is an activity index that measures disease activity and records feature of active lupus as present or not present. SLEDAI-2K uses a weighted checklist to assign a numerical score based on the presence or absence of 24 symptoms. Each symptom present is assigned between 1 and 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms).
Time Frame: Baseline: Core study Screening; LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: mITT analysis set was used. For this outcome measure, baseline was measured as reference timepoint for response in the screening visit from core study. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Participants
  LTE Day 1 | 42 | 52 | 57
  LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  LTE Week 24 | 43 | 57 | 60
  LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  LTE Week 48 | 44 | 46 | 51
  LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  LTE Week 72 | 21 | 23 | 23
  LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  LTE Week 96 | 6 | 9 | 12

9. Secondary Outcome: Number of Participants Who Achieved BILAG-based Combined Lupus Assessment (BICLA) Response (a Disease Activity Composite Index)
Description: The BICLA response was defined as BILAG-2004 improvement (all screening visit BILAG A improving to B/C/D, all screening visit BILAG B to C/D, and less than or equal to (<=1) new BILAG B and no new BILAG A); no deterioration in SLEDAI total score; PGA increase by less than (<) 0 percentage (%) (defined as less then (<)0.3 point increase for the statistical analyses) and no non-permitted medication/treatment. Baseline was defined as core study screening visit.
Time Frame: Baseline: Core study Screening; LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: mITT BILAG analysis set included mITT population with at least one BILAG A and/or B at screening visit. Here "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 76 | 70 | 86
Participants
  LTE Day 1 | 43 | 43 | 50
  LTE Week 24: number analyzed (Participants) | 67 | 66 | 81
  LTE Week 24 | 40 | 45 | 53
  LTE Week 48: number analyzed (Participants) | 55 | 55 | 68
  LTE Week 48 | 35 | 34 | 43
  LTE Week 72: number analyzed (Participants) | 29 | 27 | 30
  LTE Week 72 | 16 | 17 | 21
  LTE Week 96: number analyzed (Participants) | 8 | 12 | 12
  LTE Week 96 | 4 | 7 | 9

10. Secondary Outcome: Percent Change From Baseline in Prednisone-equivalent Corticosteroid Dose
Time Frame: Baseline: Screening Visit (Core Study); LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Percent change
  Percent Change at LTE Day 1: number analyzed (Participants) | 83 | 82 | 87
  Percent Change at LTE Day 1 | -11.04 (31.139) | -5.25 (55.697) | -11.54 (26.117)
  Percent Change at LTE Week 24: number analyzed (Participants) | 73 | 74 | 83
  Percent Change at LTE Week 24 | -11.89 (41.411) | -4.79 (59.371) | -1.21 (94.677)
  Percent Change at LTE Week 48: number analyzed (Participants) | 61 | 62 | 69
  Percent Change at LTE Week 48 | -9.19 (54.364) | -6.01 (45.605) | -17.97 (37.040)
  Percent Change at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Percent Change at LTE Week 72 | -19.32 (38.157) | -8.69 (28.112) | -22.34 (36.058)
  Percent Change at LTE Week 96: number analyzed (Participants) | 15 | 17 | 14
  Percent Change at LTE Week 96 | -36.67 (58.146) | -12.40 (73.793) | -28.57 (43.080)

11. Secondary Outcome: Change From Baseline in the Short-Form (SF-36) Health Survey Physical Component Score and Mental Component Score
Description: The 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being. These eight subscales were summarized as relating to either physical health or mental health. Physical component summary (PCS) is based primarily on physical functioning, role-physical, bodily pain, and general health scales and mental component summary (MCS) encompasses vitality, social functioning, role-emotional, and mental health scales. Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0-100 (100=highest level of mental functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100=highest level of physical functioning).
Time Frame: Baseline (Core Study Day 1); LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  PCS: Baseline (Core Study Day 1): number analyzed (Participants) | 81 | 81 | 85
  PCS: Baseline (Core Study Day 1) | 37.7 (9.20) | 37.8 (10.56) | 38.8 (9.27)
  PCS: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 85
  PCS: Change at LTE Day 1 | 4.8 (10.00) | 4.8 (8.30) | 4.0 (7.46)
  PCS: Change at LTE Week 24: number analyzed (Participants) | 72 | 74 | 80
  PCS: Change at LTE Week 24 | 5.3 (8.62) | 5.1 (8.78) | 5.9 (7.74)
  PCS: Change at LTE Week 48: number analyzed (Participants) | 59 | 61 | 66
  PCS: Change at LTE Week 48 | 6.4 (9.56) | 6.2 (9.67) | 4.6 (8.23)
  PCS: Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  PCS: Change at LTE Week 72 | 5.8 (8.61) | 3.4 (7.37) | 6.7 (5.33)
  PCS: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  PCS: Change at LTE Week 96 | 13.0 (9.51) | 3.1 (9.29) | 8.9 (6.08)
  MCS: Baseline (Core Study Day 1): number analyzed (Participants) | 81 | 81 | 85
  MCS: Baseline (Core Study Day 1) | 41.3 (10.70) | 43.3 (12.09) | 43.2 (10.81)
  MCS: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 85
  MCS: Change at LTE Day 1 | 2.1 (11.38) | 2.2 (12.62) | 1.9 (9.30)
  MCS: Change at LTE Week 24: number analyzed (Participants) | 72 | 74 | 80
  MCS: Change at LTE Week 24 | 4.4 (10.43) | 3.0 (11.75) | 2.0 (10.26)
  MCS: Change at LTE Week 48: number analyzed (Participants) | 59 | 61 | 66
  MCS: Change at LTE Week 48 | 3.3 (11.72) | 2.8 (13.19) | 3.5 (11.39)
  MCS Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  MCS Change at LTE Week 72 | 3.8 (10.96) | 1.1 (11.74) | 1.5 (13.64)
  MCS: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  MCS: Change at LTE Week 96 | 10.3 (15.86) | 0.6 (9.03) | 3.2 (12.20)

12. Secondary Outcome: Change From Baseline in Lupus Quality of Life (LupusQoL) Questionnaire Score
Description: The LupusQoL was a lupus-specific health related QoL (HRQoL) questionnaire consisting of 34 items grouped in 8 domains: physical health, pain, planning, intimate relationships, burden to others, emotional health, body image, and fatigue. Participants indicate their responses on a 5-point Likert response format, where 4 = never, 3 = occasionally, 2 = a good bit of the time, 1 = most of the time, and 0 = all of the time. Summary scores can be calculated for all 8 domains. A LupusQoL score for each domain was reported on a 0 to 100 scale, with greater values indicating better HRQoL. Baseline was defined as Day 1 of core study.
Time Frame: Baseline (Core Study Day 1); LTE Day 1, Week 24, Week 48, Week 72, and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Physical Health: Baseline (Core study Day 1): number analyzed (Participants) | 81 | 82 | 86
  Physical Health: Baseline (Core study Day 1) | 60.2 (23.08) | 62.0 (27.17) | 61.3 (27.87)
  Physical Health: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 86
  Physical Health: Change at LTE Day 1 | 8.8 (21.86) | 7.5 (17.37) | 8.2 (16.40)
  Physical Health: Change at LTE Week 24: number analyzed (Participants) | 72 | 75 | 81
  Physical Health: Change at LTE Week 24 | 10.4 (21.27) | 10.8 (18.86) | 10.9 (18.46)
  Physical Health: Change at LTE Week 48: number analyzed (Participants) | 58 | 62 | 67
  Physical Health: Change at LTE Week 48 | 9.3 (22.23) | 11.2 (24.80) | 12.8 (20.30)
  Physical Health: Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Physical Health: Change at LTE Week 72 | 8.0 (19.42) | 5.9 (17.61) | 11.9 (20.02)
  Physical Health: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Physical Health: Change at LTE Week 96 | 25.0 (21.46) | 12.9 (17.97) | 14.4 (10.33)
  Pain: Baseline (Core study Day 1): number analyzed (Participants) | 81 | 82 | 86
  Pain: Baseline (Core study Day 1) | 58.7 (26.77) | 61.2 (30.27) | 57.7 (31.52)
  Pain: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 86
  Pain: Change at LTE Day 1 | 11.8 (24.86) | 11.0 (23.93) | 13.4 (21.78)
  Pain: Change at LTE Week 24: number analyzed (Participants) | 72 | 75 | 81
  Pain: Change at LTE Week 24 | 14.4 (26.21) | 11.9 (23.38) | 16.4 (24.10)
  Pain: Change at LTE Week 48: number analyzed (Participants) | 58 | 62 | 67
  Pain: Change at LTE Week 48 | 12.8 (27.76) | 14.0 (29.64) | 17.3 (24.67)
  Pain: Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Pain: Change at LTE Week 72 | 16.7 (26.73) | 10.3 (18.91) | 17.2 (26.63)
  Pain: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Pain: Change at LTE Week 96 | 41.7 (30.21) | 11.9 (23.73) | 17.9 (23.78)
  Planning: Baseline (Core study Day 1): number analyzed (Participants) | 81 | 82 | 86
  Planning: Baseline (Core study Day 1) | 65.6 (27.52) | 68.3 (30.81) | 64.6 (33.26)
  Planning: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 86
  Planning: Change at LTE Day 1 | 8.4 (25.60) | 1.5 (22.79) | 7.5 (23.08)
  Planning: Change at LTE Week 24: number analyzed (Participants) | 72 | 75 | 81
  Planning: Change at LTE Week 24 | 11.2 (27.34) | 7.0 (24.16) | 8.4 (25.29)
  Planning: Change at LTE Week 48: number analyzed (Participants) | 58 | 62 | 67
  Planning: Change at LTE Week 48 | 14.5 (29.27) | 6.5 (26.88) | 10.9 (26.16)
  Planning: Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Planning: Change at LTE Week 72 | 10.3 (22.23) | 0.0 (28.37) | 15.5 (30.52)
  Planning: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Planning: Change at LTE Week 96 | 19.8 (36.98) | 3.0 (24.59) | 21.8 (26.03)
  Intimate Relationship: Baseline (Core study Day 1): number analyzed (Participants) | 67 | 74 | 66
  Intimate Relationship: Baseline (Core study Day 1) | 67.2 (30.99) | 60.6 (34.17) | 62.1 (31.62)
  Intimate Relationship: Change at LTE Day 1: number analyzed (Participants) | 57 | 64 | 55
  Intimate Relationship: Change at LTE Day 1 | 3.9 (26.95) | 0.2 (27.77) | -1.6 (23.94)
  Intimate Relationship: Change at LTE Week 24: number analyzed (Participants) | 48 | 60 | 52
  Intimate Relationship: Change at LTE Week 24 | 3.6 (26.29) | 7.1 (24.50) | 6.3 (25.67)
  Intimate Relationship: Change at LTE Week 48: number analyzed (Participants) | 38 | 48 | 43
  Intimate Relationship: Change at LTE Week 48 | 2.3 (29.19) | 5.7 (33.02) | 8.4 (30.58)
  Intimate Relationship: Change at LTE Week 72: number analyzed (Participants) | 18 | 27 | 24
  Intimate Relationship: Change at LTE Week 72 | -6.3 (20.67) | -2.8 (29.89) | 5.2 (32.95)
  Intimate Relationship: Change at LTE Week 96: number analyzed (Participants) | 5 | 13 | 7
  Intimate Relationship: Change at LTE Week 96 | 12.5 (15.31) | 2.9 (16.26) | -14.3 (39.81)
  Burden to Others: Baseline (Core study Day 1): number analyzed (Participants) | 81 | 82 | 86
  Burden to Others: Baseline (Core study Day 1) | 49.0 (31.22) | 48.5 (32.34) | 47.3 (32.97)
  Burden to Others: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 86
  Burden to Others: Change at LTE Day 1 | 13.4 (26.31) | 14.7 (25.83) | 12.5 (25.36)
  Burden to Others: Change at LTE Week 24: number analyzed (Participants) | 72 | 75 | 81
  Burden to Others: Change at LTE Week 24 | 13.1 (26.08) | 16.8 (27.35) | 15.7 (27.73)
  Burden to Others: Change at LTE Week 48: number analyzed (Participants) | 58 | 62 | 67
  Burden to Others: Change at LTE Week 48 | 13.4 (25.69) | 18.3 (30.36) | 17.9 (28.73)
  Burden to Others: Change at Week 72: number analyzed (Participants) | 29 | 30 | 29
  Burden to Others: Change at Week 72 | 12.1 (21.89) | 14.4 (32.23) | 22.1 (31.68)
  Burden to Others: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Burden to Others: Change at LTE Week 96 | 17.7 (32.56) | 20.2 (33.29) | 30.1 (37.51)
  Emotional Health: Baseline (Core study Day 1): number analyzed (Participants) | 81 | 82 | 86
  Emotional Health: Baseline (Core study Day 1) | 64.1 (23.43) | 68.3 (25.86) | 67.6 (27.10)
  Emotional Health: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 86
  Emotional Health: Change at LTE Day 1 | 7.9 (19.73) | 6.0 (20.08) | 7.0 (21.21)
  Emotional Health: Change at LTE Week 24: number analyzed (Participants) | 72 | 75 | 81
  Emotional Health: Change at LTE Week 24 | 11.2 (20.67) | 6.7 (21.87) | 7.9 (20.68)
  Emotional Health: Change at LTE Week 48: number analyzed (Participants) | 58 | 62 | 67
  Emotional Health: Change at LTE Week 48 | 14.2 (21.91) | 9.3 (25.66) | 8.0 (21.73)
  Emotional Health: Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Emotional Health: Change at LTE Week 72 | 10.1 (20.49) | 3.2 (17.50) | 11.5 (26.30)
  Emotional Health: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Emotional Health: Change at LTE Week 96 | 22.4 (26.16) | 6.8 (12.40) | 16.3 (22.08)
  Body Image: Baseline (Core study Day 1): number analyzed (Participants) | 76 | 71 | 82
  Body Image: Baseline (Core study Day 1) | 63.8 (27.82) | 61.9 (31.45) | 64.4 (30.51)
  Body Image: Change at LTE Day 1: number analyzed (Participants) | 61 | 67 | 72
  Body Image: Change at LTE Day 1 | 12.9 (24.47) | 6.2 (20.69) | 4.7 (25.29)
  Body Image: Change at LTE Week 24: number analyzed (Participants) | 59 | 60 | 64
  Body Image: Change at LTE Week 24 | 13.2 (25.94) | 9.1 (22.33) | 4.5 (29.34)
  Body Image: Change at LTE Week 48: number analyzed (Participants) | 45 | 54 | 55
  Body Image: Change at LTE Week 48 | 11.6 (25.39) | 14.9 (25.10) | 7.5 (28.45)
  Body Image: Change at Week 72: number analyzed (Participants) | 22 | 28 | 22
  Body Image: Change at Week 72 | 11.0 (19.15) | 8.5 (16.34) | 13.8 (29.79)
  Body Image: Change at LTE Week 96: number analyzed (Participants) | 8 | 13 | 10
  Body Image: Change at LTE Week 96 | 27.1 (32.79) | 13.4 (21.87) | 10.5 (38.19)
  Fatigue: Baseline (Core study Day 1): number analyzed (Participants) | 81 | 82 | 86
  Fatigue: Baseline (Core study Day 1) | 53.4 (26.83) | 55.6 (27.82) | 56.8 (29.00)
  Fatigue: Change at LTE Day 1: number analyzed (Participants) | 81 | 81 | 86
  Fatigue: Change at LTE Day 1 | 9.3 (21.47) | 5.9 (21.05) | 7.0 (20.93)
  Fatigue: Change at LTE Week 24: number analyzed (Participants) | 72 | 75 | 81
  Fatigue: Change at LTE Week 24 | 10.6 (23.77) | 7.1 (20.89) | 8.2 (21.96)
  Fatigue: Change at LTE Week 48: number analyzed (Participants) | 58 | 62 | 67
  Fatigue: Change at LTE Week 48 | 7.1 (23.28) | 11.9 (22.05) | 10.8 (20.05)
  Fatigue: Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Fatigue: Change at LTE Week 72 | 6.7 (25.98) | 2.7 (20.55) | 14.7 (30.63)
  Fatigue: Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Fatigue: Change at LTE Week 96 | 21.1 (33.73) | 2.7 (23.09) | 20.2 (21.06)

13. Secondary Outcome: Number of Participants With Patient Global Impression of Change (PGIC)
Description: The PGIC is self-rated scale that asks the participant to describe the change in activity limitations, symptoms, emotions, and overall Quality of life (QoL) related to the participant's painful condition on the following scale: 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) and 7 (very much worse). Number of participants in the PGIC categories of very much improved (1) and much improved (2) are reported.
Time Frame: Baseline (Core Study Day 1); LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Participants
  LTE Day 1: Very much improved | 13 | 19 | 25
  LTE Day 1: Much improved | 29 | 33 | 27
  LTE Week 24: Very much improved: number analyzed (Participants) | 74 | 75 | 83
  LTE Week 24: Very much improved | 18 | 22 | 22
  LTE Week 24: Much improved: number analyzed (Participants) | 74 | 75 | 83
  LTE Week 24: Much improved | 35 | 29 | 40
  LTE Week 48: Very much improved: number analyzed (Participants) | 61 | 63 | 70
  LTE Week 48: Very much improved | 16 | 20 | 24
  LTE Week 48: Much improved: number analyzed (Participants) | 61 | 63 | 70
  LTE Week 48: Much improved | 26 | 24 | 30
  LTE Week 72: Very much improved: number analyzed (Participants) | 33 | 30 | 32
  LTE Week 72: Very much improved | 7 | 10 | 10
  LTE Week 72: Much improved: number analyzed (Participants) | 33 | 30 | 32
  LTE Week 72: Much improved | 13 | 13 | 13
  LTE Week 96: Very much improved: number analyzed (Participants) | 9 | 14 | 13
  LTE Week 96: Very much improved | 4 | 2 | 7
  LTE Week 96: Much improved: number analyzed (Participants) | 9 | 14 | 13
  LTE Week 96: Much improved | 4 | 7 | 5

14. Secondary Outcome: Change From Baseline in EuroQoL 5 Dimension Instrument (EQ-5D) Score
Description: EQ-5D questionnaire comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression measured on 3 levels; 1=no problem, 2=moderate problems, 3=extreme problems. This part, called the EQ-5D descriptive system, provides a 5-dimensional description of health status. 5 dimensional 3-level system was converted into single index utility score. Possible values for single index utility score ranged from -0.594 (severe problems in all dimensions) to 1.0 (no problem in all dimensions) on scale where 1 represented best possible health state. Baseline was defined as Day 1 of Core study.
Time Frame: Baseline: Day 1 (Core Study), LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Baseline (Core Study Day 1): number analyzed (Participants) | 82 | 82 | 86
  Baseline (Core Study Day 1) | 0.736 (0.1707) | 0.775 (0.1754) | 0.751 (0.2388)
  Change at LTE Day 1: number analyzed (Participants) | 82 | 82 | 86
  Change at LTE Day 1 | 0.038 (0.1764) | 0.042 (0.1759) | 0.070 (0.1912)
  Change at LTE Week 24: number analyzed (Participants) | 73 | 75 | 81
  Change at LTE Week 24 | 0.078 (0.1651) | 0.024 (0.2207) | 0.072 (0.1933)
  Change at LTE Week 48: number analyzed (Participants) | 59 | 62 | 67
  Change at LTE Week 48 | 0.065 (0.2050) | 0.045 (0.2393) | 0.076 (0.2414)
  Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Change at LTE Week 72 | 0.045 (0.1531) | 0.000 (0.2126) | 0.087 (0.2609)
  Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Change at LTE Week 96 | 0.138 (0.1257) | -0.015 (0.1767) | 0.132 (0.1927)

15. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS) Scores
Description: EQ-5D is a participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeters (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state. Baseline defined as Day 1 of core study.
Time Frame: Baseline: Day 1 (Core Study), LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
mm
  Baseline (Core Study Day 1): number analyzed (Participants) | 82 | 82 | 85
  Baseline (Core Study Day 1) | 61 (18.8) | 65 (21.4) | 65 (22.2)
  Change at LTE Day 1: number analyzed (Participants) | 82 | 82 | 85
  Change at LTE Day 1 | 9 (16.0) | 11 (21.5) | 8 (18.1)
  Change at LTE Week 24: number analyzed (Participants) | 73 | 75 | 80
  Change at LTE Week 24 | 13 (19.7) | 12 (21.4) | 11 (18.4)
  Change at LTE Week 48: number analyzed (Participants) | 59 | 62 | 66
  Change at LTE Week 48 | 15 (18.4) | 14 (23.9) | 9 (19.6)
  Change at LTE Week 72: number analyzed (Participants) | 29 | 30 | 29
  Change at LTE Week 72 | 12 (18.9) | 12 (19.6) | 10 (18.1)
  Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Change at LTE Week 96 | 19 (17.6) | 12 (20.9) | 10 (21.6)

16. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. It uses a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse possible score) to 52 (best score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline: Day 1 (Core study); LTE Day 1, Week 24, Week 48, Week 72 and Week 96
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Units on a scale
  Baseline; Day 1 (Core Study): number analyzed (Participants) | 81 | 81 | 86
  Baseline; Day 1 (Core Study) | 29 (10.1) | 32 (13.1) | 31 (13.1)
  Change at LTE Day 1: number analyzed (Participants) | 81 | 80 | 86
  Change at LTE Day 1 | 4 (9.5) | 4 (10.2) | 4 (9.8)
  Change at LTE Week 24: number analyzed (Participants) | 72 | 74 | 81
  Change at LTE Week 24 | 5 (10.1) | 3 (10.9) | 4 (9.9)
  Change at LTE Week 48: number analyzed (Participants) | 58 | 61 | 67
  Change at LTE Week 48 | 5 (11.2) | 4 (12.3) | 5 (9.9)
  Change at LTE Week 72: number analyzed (Participants) | 29 | 29 | 29
  Change at LTE Week 72 | 4 (11.3) | 2 (10.2) | 6 (10.2)
  Change at LTE Week 96: number analyzed (Participants) | 8 | 14 | 13
  Change at LTE Week 96 | 13 (15.5) | 3 (8.4) | 9 (9.2)

17. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. Treatment-Emergent adverse events (TEAEs) are defined as events with an onset date on or after the date of first dose of study treatment in the core study and ongoing at LTE study entry, or occurring during LTE study.
Time Frame: Baseline (Day 1 of Core study) up to maximum duration of 167.7 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Participants | 68 | 67 | 76

18. Secondary Outcome: Number of Participants With Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: The C-SSRS assesses the suicidal behavior and suicidal ideation in participants. Occurrence of suicidal behavior after study entry is defined as having answered "yes" to a least 1 of the 4 suicidal behavior subcategories (actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior). Occurrence of suicidal ideation is defined as having answered "yes" to at least 1 of the suicidal ideation sub-categories (1) wish to be dead, (2) nonspecific active suicidal thoughts, (3) active suicidal ideation with any methods (no plan) without intent to act, (4) active suicidal ideation with some intent to act (without specific plan), and (5) active suicidal ideation with specific plan and intent).
Time Frame: LTE Day 1, Week 24, Week 48, Week 72 and Week 98
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 83 | 82 | 88
Participants
  Occurrence of Suicidal Behavior at LTE Day 1 | 0 | 0 | 0
  Occurrence of Suicidal Behavior at LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  Occurrence of Suicidal Behavior at LTE Week 24 | 0 | 0 | 0
  Occurrence of Suicidal Behavior at LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  Occurrence of Suicidal Behavior at LTE Week 48 | 0 | 0 | 0
  Occurrence of Suicidal Behavior at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Occurrence of Suicidal Behavior at LTE Week 72 | 0 | 0 | 0
  Occurrence of Suicidal Behavior at LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  Occurrence of Suicidal Behavior at LTE Week 96 | 0 | 0 | 0
  Occurrence of Suicidal Ideation at LTE Day 1 | 0 | 0 | 0
  Occurrence of Suicidal Ideation at LTE Week 24: number analyzed (Participants) | 74 | 75 | 83
  Occurrence of Suicidal Ideation at LTE Week 24 | 0 | 0 | 0
  Occurrence of Suicidal Ideation at LTE Week 48: number analyzed (Participants) | 61 | 63 | 70
  Occurrence of Suicidal Ideation at LTE Week 48 | 0 | 0 | 0
  Occurrence of Suicidal Ideation at LTE Week 72: number analyzed (Participants) | 33 | 30 | 32
  Occurrence of Suicidal Ideation at LTE Week 72 | 1 | 0 | 1
  Occurrence of Suicidal Ideation at LTE Week 96: number analyzed (Participants) | 9 | 14 | 13
  Occurrence of Suicidal Ideation at LTE Week 96 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to maximum duration of 167.7 weeks
Description: The safety analyses set included all participants enrolled into the LTE study and who received at least 1 dose of planned study treatment. Participants were analyzed according to the actual treatment they received.
Arm/Group | Placebo/Atacicept 150 mg | Atacicept 75 mg | Atacicept 150 mg
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/82 | 2/88
Serious Adverse Events (participants affected / at risk) | 19/83 | 13/82 | 11/88
Other Adverse Events (participants affected / at risk) | 65/83 | 65/82 | 75/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Atacicept 150 mg (N=83) | Atacicept 75 mg (N=82) | Atacicept 150 mg (N=88)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Embryonal rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 0 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system lupus (Nervous system disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Atacicept 150 mg (N=83) | Atacicept 75 mg (N=82) | Atacicept 150 mg (N=88)
Urinary tract infection (Infections and infestations) | 18 | 14 | 17
Upper respiratory tract infection (Infections and infestations) | 7 | 11 | 15
Nasopharyngitis (Infections and infestations) | 8 | 8 | 5
Bronchitis (Infections and infestations) | 7 | 10 | 2
Sinusitis (Infections and infestations) | 3 | 7 | 5
Pharyngitis (Infections and infestations) | 3 | 6 | 6
Injection site reaction (General disorders) | 23 | 14 | 22
Injection site pain (General disorders) | 11 | 4 | 14
Injection site erythema (General disorders) | 5 | 3 | 1
Gastritis (Gastrointestinal disorders) | 5 | 2 | 4
Headache (Nervous system disorders) | 11 | 3 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 4
Hypertension (Vascular disorders) | 1 | 4 | 6

LIMITATIONS AND CAVEATS:
The study was terminated early due to shortage of drug supply and there were many fewer number of participants remaining in each dosage group after Week 72 preluding meaningful inferences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes